CLINICAL TRIAL: NCT01173237
Title: Efficacy Evaluation of Surfactant Administration for Respiratory Distress Syndrome Treatment Via Laryngeal Mask Airway. A Randomized Controlled Trial
Brief Title: Efficacy Evaluation of Surfactant Administration Via Laryngeal Mask Airway
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Rosilu Ferreira Barbosa, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE 00160287000-10
Record Dates: First submitted 2010-07-26; First posted 2010-08-02 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2010-07

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: tracheal intubation; proseal laryngeal mask airway; neonate; surfactant; respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Respiratory Distress Syndrome | interventions — Laryngeal Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tracheal intubation (Active Comparator): Endotracheal tube is a airway device used for ventilation or surfactant administration, in preterm babies with SDR surfactant deficiency.
  Interventions: Procedure: Use tracheal intubation for surfactant therapy
- Proseal laryngeal mask airway (Experimental): Laryngeal mask airway is a airway device used for ventilation with self-inflating bag or flow-inflating bag. In this study it will be used for surfactant administration, in preterm babies with SDR surfactant deficiency.
  Interventions: Procedure: Use of Proseal laryngeal mask airway for surfactant therapy

INTERVENTIONS:
Procedure: Use tracheal intubation for surfactant therapy — Surfactant endotracheal administration after tracheal intubation
  Other Names: Endotracheal tube
  Arms: Tracheal intubation
Procedure: Use of Proseal laryngeal mask airway for surfactant therapy — Surfactant use by proseal laryngeal mask airway
  Other Names: Laryngeal mask airway
  Arms: Proseal laryngeal mask airway

SUMMARY:
With the development of the Intubation Surfactant Extubation technic, in which surfactant is administered during a brief intubation followed by immediate extubation, surfactant therapy can be given during nasal continuous positive airway pressure treatment further reducing need for mechanical ventilation. Preterm newborn babies until eight hours of life, with respiratory distress syndrome, will be randomized to standard delivery of surfactant via endotracheal tube airway inserted after premedication for pain with midazolam and remifentanil or to surfactant delivery via Proseal laryngeal mask airway size 1. The intent is to is to compare efficacy and safety of surfactant administration via two different airways and ventilatory approaches.

ELIGIBILITY:
Inclusion Criteria:

* Birthweight more than 1000 grams
* Gestational age more than 28 weeks and less than 35 weeks
* Chronologic age less than 8 hours
* Diagnosis of RDS by clinical and radiographic criteria
* Treated with nasal continuous positive airway pressure and supplemental oxygen more than 30%
* Parental consent

Exclusion Criteria:

* Birthweight less than 1000 grams
* Gestational age more than 28 weeks and less than 35 weeks
* Chronologic age more than 8 hours
* Maternal fever or premature rupture of fetal membranes less than 18 hours
* Diagnosis other than respiratory distress syndrome
* Babies who require or have already had endotracheal intubation
* Analgesia and or sedation during the first six hours of life
* Apgar 5 minute score less than three
* Babies with congenital anomalies or signs of acute circulatory failure

Ages: 30 Minutes to 8 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-03 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Fraction of inspired oxygen | three hours

SECONDARY OUTCOMES:
Hormonal evaluation of pain | three hours
Proseal laryngeal mask surfactant treatment failure | Six hours
Rate of respiratory distress syndrome complications | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Yerkes P Silva, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (2):
- Brazil (2):
  - Maternidade Odete Valadares, Belo Horizonte, Minas Gerais
  - Hospital Dia e Maternidade Unimed-BH, Belo Horizonte, Minas Gerais